CLINICAL TRIAL: NCT06750575
Title: The Effect of Furosemide on Protein-Bound Uremic Toxin Plasma Levels and Excretion in Patients with Chronic Kidney Disease
Brief Title: Study to Examine the Effect of the Diuretic Furosemide on the Plasma Levels of Toxins and the Removal of Toxins from the Blood in Patients with Chronic Kidney Disease
Acronym: FUROPBUT
Status: Recruiting | Type: Observational
Sponsor: UMC Utrecht (Other)
Collaborators: Maastricht University, MERLN Institute for Technology-Inspired Regenerative Medicine (Unknown); Utrecht Institute for Pharmaceutical Sciences (Other)
Responsible Party: Principal Investigator, Karin G.F. Gerritsen, Associate professor, MD, UMC Utrecht
Other Study IDs: NL81338.041.23; 23-239/G (Other: Medical Ethics Committee NedMec)
Record Dates: First submitted 2024-10-17; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Chronic Kidney Diseases; Renal Failure Chronic
Keywords: Furosemide; Drug-toxin interactions; Protein-bound uremic toxins; P-cresyl sulfate; Indoxyl sulfate
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and urine samples will be temporarily retained during this study for batch measurement. Afterwards, the samples will be retained until publication of the data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Chronic kidney disease stage 3-5: Participants with an age of 18 years or older and with CKD stage 3-5 (an estimated glomerular filtration rate of 60 mL/min/1.73m^2 or lower for at least three months). Participants need to have an indication to start with furosemide as part of routine patient care.
  Interventions: Diagnostic Test: Invasive measurements

INTERVENTIONS:
Diagnostic Test: Invasive measurements — Blood and urine samples will be collected during the study.

SUMMARY:
The goal of this observational study is to examine the interaction between the diuretic furosemide and certain toxins called protein-bound uremic toxins (PBUTs) in patients with chronic kidney disease (CKD). The main question it aims to answer is: what is the effect of furosemide on plasma levels of PBUTs in patients with CKD? Besides, the investigators will also look at the effect of furosemide on the excretion of PBUTs via the urine.

Participants will be included in the study once they will be prescribed furosemide as part of routine patient care. Before they start with the furosemide treatment, patients will undergo the following:

* Blood pressure measurement
* Blood sample withdrawal
* Urine sample collection
* 12-hour urine collection

Then, one to four weeks after starting with furosemide treatment, patients will undergo the following:

* Blood pressure measurement
* Blood sample prior to furosemide intake (Tmin)
* Blood sample withdrawal 90 minutes after furosemide intake (Tmax: time at which the highest furosemide plasma level is expected)
* Urine sample collection 60-120 minutes after furosemide intake
* 12-hour urine collection

The investigators expect furosemide to increase plasma levels of PBUTs by decreasing the renal excretion of the toxins.

DETAILED DESCRIPTION:
Protein-bound uremic toxins are known to accumulate in chronic kidney disease (CKD) and are associated with increased morbidity and mortality. It is therefore crucial to maintain the PBUT levels low in this patient group. Furosemide is often prescribed to CKD patients. However, based on preclinical data, furosemide could affect the renal excretion of PBUTs, either by competing for binding to albumin or by competing for the secretory system in the kidney. It is important to examine the effect of furosemide on the excretion and plasma concentration PBUTs as this might have harmful consequences for patients with CKD.

This study aims to examine the effect of furosemide PBUT plasma levels in patients with CKD as well as the renal PBUT excretion. The investigators expect furosemide to increase plasma levels of PBUTs by decreasing the renal excretion of the toxins.

This study is observational and includes invasive measurements; a prospective repeated measures cohort study design will be used in which PBUT plasma concentrations and excretion will be determined before and after the start of furosemide treatment.

The study population consists of patients with CKD stage 3-5 (<60 mL/min/1.73m2 for at least three months) who have an indication for furosemide treatment as part of routine patient care. Participants will receive furosemide in a dosage prescribed by their nephrologist as part of their routine patient care; this treatment is not changed by the participation of patients in the study.

A power analysis for a paired samples T-Test was done using GPower (version 3.1.9.4). Data regarding PBUT plasma levels from the study of Tang et al. in 2021 was used in order to calculate the sample size; PCS plasma levels before (average ± standard deviation: 13,481 ± 12,642 nM) and after (average ± standard deviation: 23,000 ± 24,900 nM) furosemide intake were chosen, since PCS is one of the main PBUTs of interest. This calculation showed a required sample size of 34 (one-tail, power = 80%, α = 0.05, d = 0.44, correlation between samples 0.5 based on assumption).

Prior to the start of the furosemide treatment, a blood sample (three tubes/11 mL per withdrawal) and a urine sample will be collected from patients enrolled in the study. Participants will also hand in a 12-hour urine collection and their blood pressure will be measured.

After the start of the furosemide treatment (at least one week after the start of the furosemide treatment so that steady state has been reached), two blood samples, one urine sample, and a 24-hour urine collection will be obtained. Participants will be asked to obtain a 12-hour urine collection and to bring this with them on the day the of the visit. During the visit at the University Medical Center Utrecht, participants will first hand in the 12-hour urine collection and their blood pressure will be measured. Furthermore, a blood sample will be taken prior to the furosemide intake (Tmin). Then, they will take their prescribed furosemide at around the same time as they normally take their medication. 60 minutes after the furosemide intake, participants will be asked to empty their bladder and drink two glasses of water. Then, at Tmax, a blood sample will be collected. Tmax is estimated at around 90 minutes after oral intake; therefore, the target time of sample collection is 90 min with an acceptable range between 60-120 minutes after furosemide intake. Furthermore, a urine sample will be collected between 60 and 120 minutes after furosemide intake in order to best examine the effect of furosemide on PBUT excretion. The exact time of furosemide intake and the time of the blood and urine sample collection will be registered.

The main endpoints of this study are PBUT plasma levels before and 1-4 weeks after the start of furosemide treatment (in a steady state).

Baseline characteristics and study parameters will be presented as either a mean with standard deviation or a median with interquartile range for continuous data, or as a percentage for categorical data. Results with a p<0.05 will be considered statistically significant. Analyses will be done using the statistical software platforms SPSS and R. Missing data will be excluded from the analyses via pairwise deletion.

Participants will only receive furosemide prescribed by their treating nephrologist as part of routine patient care. In addition, three blood sample drawings, two urine samples, and two 12-hour urine collections will be needed. Thus, the risk associated with participation is negligibly low. Participation to the study will include two site visits. These visits will be combined with routine check-ups as much as possible.

ELIGIBILITY:
Inclusion Criteria:

* An age of 18 years or older
* An eGFR <60 mL/min/1.73m2 for at least three months (diagnosis of CKD stage 3-5)
* An indication for the start of treatment with furosemide as part of routine patient care
* Willingness to participate in the study and a signed informed consent

Exclusion Criteria:

* Patients who are already on furosemide treatment
* Patients with a liver disease with hyperbilirubinemia
* Patients who receive any type of renal replacement therapy (peritoneal dialysis, haemodialysis)
* Patients with end-stage renal failure without residual diuresis
* Patients who will start with medication simultaneously with start of furosemide treatment that might interfere with PBUT excretion or PBUT protein binding
* Patients who are incapacitated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients with CKD stage 3-5 (eGFR <60 mL/min/1.73m2) of 18 years and older with an indication for starting treatment with furosemide as part of routine patient care. Participants will be recruited at the Department of Nephrology in the University Medical Center Utrecht (UMCU, Utrecht, The Netherlands) who have not yet started furosemide treatment or any renal replacement therapy.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Plasma levels of the PBUT indoxyl sulfate | This will be assessed three times during the study participation period (between 1-4 weeks).
  Indoxyl sulfate plasma levels (in ng/mL) will be determined before and after start of furosemide treatment.
Plasma levels of the PBUT p-cresyl sulfate | This will be assessed three time during the study participation period (between 1-4 weeks).
  P-cresyl sulfate plasma levels (in ng/mL) will be determined before and after start of furosemide treatment.
Plasma levels of the PBUT indole-3-acetic acid | This will be assessed three times during the study participation period (between 1-4 weeks).
  Indole-3-acetic acid plasma levels (in ng/mL) will be determined before and after start of furosemide treatment.
Plasma levels of the PBUT kynurenic acid | This will be assessed three times during the study participation period (between 1-4 weeks).
  Kynurenic acid plasma levels (in ng/mL) will be determined before and after start of furosemide treatment.
Plasma levels of the PBUT L-kynurenine | This will be assessed three times during the study participation period (between 1-4 weeks).
  L-kynurenine plasma levels (in ng/mL) will be determined before and after start of furosemide treatment.
Plasma levels of the PBUT hippuric acid | This will be assessed three times during the study participation period (between 1-4 weeks).
  Hippuric acid plasma levels (in ng/mL) will be determined before and after start of furosemide treatment.
Plasma levels of the PBUT p-cresyl glucuronide | This will be assessed three times during the study participation period (between 1-4 weeks).
  P-cresyl glucuronide plasma levels (in ng/mL) will be determined before and after start of furosemide treatment.

SECONDARY OUTCOMES:
Surrogate for PBUT clearance | This will be assessed three times during the study participation period (between 1-4 weeks).
  This will be calculated for seven PBUTs (indoxyl sulfate, p-cresyl sulfate, indole-3-acetic acid, kynurenic acid, L-kynurenine, hippuric acid, p-cresyl glucuronide) before and after start of furosemide treatment using the following formula:
  Urine PBUT concentration / (urine creatinine concentration * plasma PBUT concentration)
Fractional PBUT excretion | This will be assessed three times during the study participation period (between 1-4 weeks).
  This will be calculated for seven PBUTs (indoxyl sulfate, p-cresyl sulfate, indole-3-acetic acid, kynurenic acid, L-kynurenine, hippuric acid, p-cresyl glucuronide) before and after start of furosemide treatment using the following formula:
  (Urine PBUT concentration * plasma creatinine concentration) / (urine creatinine concentration * plasma PBUT concentration)
PBUT protein binding | This will be assessed three times during the study participation period (between 1-4 weeks).
  This will be determined for seven PBUTs (indoxyl sulfate, p-cresyl sulfate, indole-3-acetic acid, kynurenic acid, L-kynurenine, hippuric acid, p-cresyl glucuronide) before and after start of furosemide treatment by determining the total PBUT plasma concentration and the free fraction of the PBUTs.
Ratio of the surrogate PBUT clearance / CKD-EPI creatinine equation | This will be assessed three times during the study participation period (between 1-4 weeks).
  This will be calculated for seven PBUTs (indoxyl sulfate, p-cresyl sulfate, indole-3-acetic acid, kynurenic acid, L-kynurenine, hippuric acid, p-cresyl glucuronide) before and after start of furosemide treatment using the following formulas:
  For surrogate of PBUT concentration:
  Urine PBUT concentration / (urine creatinine concentration * plasma PBUT concentration)
  For CKD-EPI creatinine equation: eGFR (in mL/min/1.73m^2) = 142* Min(Scr/K, 1)^α * Max(Scr/K, 1)^-1.200 * 0.9938^Age (in years) * 1.012 [if female]
  In which:
  eGFR = estimated glomerular filtration rate Scr = serum creatinine in mg/dL K = 0.7 for females, 0.9 for males α = -0.241 for females, -0.302 for males Min(Scr/K, 1) = the minimum of Scr/K or 1 Max(Scr/K, 1) = the maximum of Scr/K or 1
Ratio of the surrogate PBUT clearance / CKD-EPI cystatin C equation | This will be assessed three times during the study participation period (between 1-4 weeks).
  This will be calculated for seven PBUTs (indoxyl sulfate, p-cresyl sulfate, indole-3-acetic acid, kynurenic acid, L-kynurenine, hippuric acid, p-cresyl glucuronide) before and after start of furosemide treatment using the following formulas:
  For surrogate of PBUT concentration:
  Urine PBUT concentration / (urine creatinine concentration * plasma PBUT concentration)
  For CKD-EPI cystatin C equation: eGFR (in mL/min/1.73m^2) = 133 * Min(Scys/0.8, 1)^-0.499 * Max(Scys/0.8, 1)^-1.328 * 0.996^Age (in years) * 0.932 [if female]
  In which:
  eGFR = estimated glomerular filtration rate Scys = serum cystatin C in mg/L Min(Scys/0.8, 1) = the minimum of Scys/0.8 or 1 Max(Scys/0.8, 1) = the maximum of Scys/0.8 or 1
Ratio of the surrogate PBUT clearance / CKD-EPI creatinine-cystatin C equation | This will be assessed three times during the study participation period (between 1-4 weeks).
  This will be calculated for seven PBUTs (indoxyl sulfate, p-cresyl sulfate, indole-3-acetic acid, kynurenic acid, L-kynurenine, hippuric acid, p-cresyl glucuronide) before and after start of furosemide treatment using the following formulas:
  For surrogate of PBUT concentration:
  Urine PBUT concentration / (urine creatinine concentration * plasma PBUT concentration)
  For CKD-EPI cystatin C equation: eGFR (in mL/min/1.73m^2) = 135 * Min(Scr/K, 1)^α * Max(Scr/K, 1)^-0.544 * Min(Scys/0.8, 1)^-0.323 * Max(Scys/0.8, 1)^-0.778 * 0.9961^Age (in years) * 0.963 [if female]
  In which:
  eGFR = estimated glomerular filtration rate Scr = serum creatinine in mg/dL Scys = serum cystatin C in mg/L K = 0.7 for females, 0.9 for males α = -0.219 for females, -0.144 for males Min(Scr/K, 1) = the minimum of Scr/K or 1 Min(Scys/0.8, 1) = the minimum of Scys/0.8 or 1 Max(Scr/K, 1) = the maximum of Scr/K or 1 Max(Scys/0.8, 1) = the maximum of Scys/0.8 or 1

OTHER OUTCOMES:
Baseline characteristics: age | This will be collected once throughout the study participation period (between 1-4 weeks) during the first study visit.
  Age (in years) will be documented during the first study visit.
Baseline characteristics: sex | This will be collected once throughout the study participation period (between 1-4 weeks) during the first study visit.
  Sex (male/female/other) will be documented during the first study visit.
Baseline characteristics: BMI | This will be collected once throughout the study participation period (between 1-4 weeks) during the first study visit.
  BMI (calculated from length and weight in kg/m^2) will be documented during the first study visit.
Prescribed dosage of furosemide | This will be collected once throughout the study participation period (between 1-4 weeks) during the first study visit.
  The prescribed dosage of furosemide (including frequency of intake and dosage per intake) will be collected during the first study visit.
Comorbidities and underlying cause of renal disease | This will be collected once throughout the study participation period (between 1-4 weeks) during the first study visit.
  Data regarding comorbidities and underlying cause of renal disease of participants will be collected during the first study visit.
Medication usage | This will be assessed twice during the study participation period (between 1-4 weeks).
  Medication usage of the participant will be assessed at both study visits.
Blood pressure measurements | This will be assessed twice during the study participation period (between 1-4 weeks).
  Blood pressure (systolic and diastolic, in mmHg) will be measured before and after start of furosemide treatment.
Postprandial or fasting state | This will be assessed twice during the study participation period (between 1-4 weeks).
  Postprandial/fasting state will be assessed at the time of blood and urine sample collection before and after start of furosemide treatment. This means that participants will be asked whether they have eaten prior to the sample collection (in the morning). If so: postprandial state. If not: fasting state.
Intake of prescribed medication | This will be assessed twice during the study participation period (between 1-4 weeks).
  Intake of prescribed medication will be assessed at the time of blood and urine sample collection before and after start of furosemide treatment.
Furosemide plasma and urine levels | This will be assessed three times in plasma and four times in urine (also in 12-hour urine collections) during the study participation period (between 1-4 weeks).
  Furosemide plasma and urine levels will be determined before and after start of furosemide treatment.
Cystatin C plasma and urine levels | This will be assessed three times in plasma and two times in urine during the study participation period (between 1-4 weeks).
  Cystatin C plasma and urine levels will be determined before and after start of furosemide treatment.
Bicarbonate plasma levels | This will be assessed three times during the study participation period (between 1-4 weeks).
  Bicarbonate plasma levels will be determined before and after start of furosemide treatment.
Neutrophil Gelatinase-Associated Lipocalin (NGAL) urine levels | This will be assessed twice during the study participation period (between 1-4 weeks).
  NGAL urine levels will be determined before and after start of furosemide treatment.
Kidney Injury Molecule-1 (KIM1) urine levels | This will be assessed twice during the study participation period (between 1-4 weeks).
  KIM1 urine levels will be determined before and after start of furosemide treatment.
Beta-2 microglobulin urine levels | This will be assessed twice during the study participation period (between 1-4 weeks).
  Beta-2 microglobulin urine levels will be determined before and after start of furosemide treatment.
Albumin plasma and urine levels | This will be assessed three times in plasma and four times in urine (also in 12-hour urine collections) during the study participation period (between 1-4 weeks).
  Albumin plasma and urine levels will be determined before and after start of furosemide treatment.
Total protein urine levels | This will be assessed four times (also in 12-hour urine collection) during the study participation period (between 1-4 weeks).
  Total protein urine levels will be determined before and after start of furosemide treatment.
Fractional urea excretion | This will be assessed twice during the study participation period (between 1-4 weeks).
  Fractional urea excretion will be calculated before and after start of furosemide treatment.
  This will be calculated using the following formula:
  (Urine urea concentration * plasma creatinine concentration) / (urine creatinine concentration * plasma urea concentration)
Urine pH | This will be assessed twice during the study participation period (between 1-4 weeks).
  Urine pH will be determined before and after start of furosemide treatment.
Furosemide protein binding | This will be assessed three times during the study participation period (between 1-4 weeks).
  This will be determined before and after start of furosemide treatment by determining the total furosemide plasma concentration and the free fraction of furosemide.
PBUT levels in the 12-hour urine collections | This will be assessed twice during the study participation period (between 1-4 weeks).
  Urine levels of seven PBUTs (indoxyl sulfate, p-cresyl sulfate, indole-3-acetic acid, kynurenic acid, L-kynurenine, hippuric acid, p-cresyl glucuronide) will be determined in the 12-hour urine collections.
Creatinine levels in the 12-hour urine collections | This will be assessed twice during the study participation period (between 1-4 weeks).
  Urine levels of creatinine will be determined in the 12-hour urine collections.
Urea levels in the 12-hour urine collections | This will be assessed twice during the study participation period (between 1-4 weeks).
  Urine levels of urea will be determined in the 12-hour urine collections.

CONTACTS AND LOCATIONS:
Overall Officials: Karin GF Gerritsen, MD, PhD, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center Utrecht (UMCU), Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The data package will contain: the raw data, the study protocol describing the methods and materials, the script to process the data, the scripts leading to tables and figures in the publication, a codebook with explanations on the variable names, and a 'read_me.txt' file with an overview of files included and their content and use.
  All data and documents in the data package will be shared under restrictions. The publication will be openly assessable. The study protocol and this Data Management Plan will also be available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Our data will be shared with third parties after approval of the Principal Investigator. The criteria and time period will be determined on a case-by-case basis.
Access Criteria: Our data will be shared with third parties after approval of the Principal Investigator. The criteria and time period will be determined on a case-by-case basis.

REFERENCES:
- [Background] Mihaila SM, Faria J, Stefens MFJ, Stamatialis D, Verhaar MC, Gerritsen KGF, Masereeuw R. Drugs Commonly Applied to Kidney Patients May Compromise Renal Tubular Uremic Toxins Excretion. Toxins (Basel). 2020 Jun 12;12(6):391. doi: 10.3390/toxins12060391. PMID 32545617